CLINICAL TRIAL: NCT06139770
Title: Treatment of Anorexia Nervosa in Children and Adolescents: An Integrated Family-based and Metacognitive Approach
Brief Title: Treatment of Anorexia Nervosa in Children and Adolescents: An Integrated Family Based and Metacognitive Approach
Acronym: FBT-MCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 255677
Record Dates: First submitted 2023-08-24; First posted 2023-11-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: The patients will receive the same treatment (FBT/MCT) including their parents, and by post treatment the patients will be randomised to two types of follow-up. One group of the patients will be allocated to active follow-up, receiving 3 booster sessions during the 12 months follow-up, and the second group will be followed-up as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active follow-up (Active Comparator): The patients will recieve 3 sessions of MCT
  Interventions: Behavioral: Family based therapy- Metacognitive therapy
- Passive follow-up (Active Comparator): The group receives no sessions during follow-up
  Interventions: Behavioral: Family based therapy- Metacognitive therapy

INTERVENTIONS:
Behavioral: Family based therapy- Metacognitive therapy — Family based therapy and Metacognitive therapy

SUMMARY:
The goal of this study is to evaluate the treatment effects of an integrated treatment called Family-based and Metacognitive therapy for patients with Anorexia Nervosa. In addition, we will evaluate if an active follow-up of the patients will reduce the number of relapses, which is common during the 1 year after discharge. Fifty patients aged 12-18 years old and their parents will be invited to participate in this study and all will receive the same treatment but be randomly allocated to different follow-up conditions. The active follow-up includes 3 sessions of Metacognitive therapy and the passive follow-up includes ordinary follow-up, with no booster sessions. The patients will be assessed at baseline, pre-treatment, post-treatment, and at 6 and 12 months follow-up.

DETAILED DESCRIPTION:
The study is an evaluation of a new approach to treating Anorexia Nervosa (F.50.0 and F 50.1) called Family-based and Metacognitive therapy. The treatment integrates both family-based work approach, where the parents learn to be in control of the meal situation and communicate better with their child. The metacognitive treatment approach, is targeting the child to work with its problems with emotional regulation and self-esteem issues, but also their attitudes to body and weight. Our aim is to both address what the overall effect of the treatment will be, but also to test if an active follow-up after discharge will lead to reduced relapse rates in the 12 months after treatment. We will apply the same approach to all included patients (A-B design), but the patients and their parents will be allocated to one of two different conditions for follow-up. The active follow-up involves receiving 3 sessions of metacognitive therapy, whereas the other group gets ordinary follow-up, with no sessions of MCT. All patients are assessed at baseline, pre-treatment, post-treatment, and by 6 and 12 months follow-up. The purpose of the design is to evaluate if the rate of relapse during the first year after discharge can be reduced

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of F 50.0 and F 50.1

Exclusion Criteria:

* Psychotic symptoms
* Severe somatic illness
* Mental retardation or developmental disorder
* Bipolar disorder
* Extreme self-mutilation or acute suicidal risks
* Does not speak or understand Norwegian

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index | 18 months
  Body mass index

CONTACTS AND LOCATIONS:
Locations (1):
- St.Olavs hospital HF, Trondheim, Trøndelag, Norway